CLINICAL TRIAL: NCT01518257
Title: Safety and Efficacy Study of Botulinum Toxin Type A as Treatment for Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-102
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- botulinum toxin Type A (Experimental): A single 200U (2 mL) dose of botulinum toxin Type A injected into the intra-articular space of the study knee on Day 1.
  Interventions: Biological: botulinum toxin Type A
- Placebo (Placebo Comparator): A single 2 mL dose of Normal Saline (placebo) injected into the intra-articular space of the study knee on Day 1.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: botulinum toxin Type A — A single 200U (2 mL) dose of botulinum toxin Type A injected into the intra-articular space of the study knee on Day 1.
  Other Names: BOTOX®
  Arms: botulinum toxin Type A
Drug: Normal Saline — A single 2 mL dose of Normal Saline (placebo) injected into the intra-articular space of the study knee on Day 1.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of a single intra-articular (IA) injection of botulinum toxin Type A compared with placebo as treatment for osteoarthritis (OA) knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Painful osteoarthritis in the study knee
* Able to walk without assistive walking devices, able to perform usual daily activities, and agree to maintain similar activity level throughout the study

Exclusion Criteria:

* Chronic pain conditions other than knee osteoarthritis
* Presence of bursitis, meniscus tear, ligament tear, or significant injury to the study knee within 1 year
* Surgery to the study knee within 24 weeks
* Treatment with hyaluronic acid in the study knee within 24 weeks
* Treatment with corticosteroids in the study knee within 12 weeks
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis
* Previous treatment with botulinum toxin of any serotype for any reason

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Aalborg, Denmark

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A | Placebo
Started | 61 | 60
Completed | 59 | 60
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other Miscellaneous Reason | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | Placebo | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Customized [Number; unit: Participants]
  40 to 64 Years | 30 | 31 | 61
  ≥ 65 Years | 31 | 29 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 62
  Male | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Daily Worst Pain Intensity Score at Week 4
Description: The patient rated their daily worst pain intensity in the study knee using an 11-point scale where: 0=no pain to 10=worst pain possible. The daily scores over the previous 14-day period were averaged. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 4
Population: Safety population included all treated participants based on the actual treatment received.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 61 | 60
Score on a scale
  Baseline | 6.4 (1.09) | 6.5 (1.28)
  Change from Baseline at Week 4 | -1.8 (1.66) | -1.8 (1.87)

2. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Arthritis (WOMAC™) Total Index Score
Description: The WOMAC Total Index Score consisted of 24 components rated on a scale of 0 to 10. The Total Index Score included the WOMAC Pain Score (5 questions about pain where: 0=no pain to 10=extreme pain), the WOMAC Physical Function score (17 questions about the difficulty of daily activities where: 0=no difficulty to 10=extreme difficulty) and the WOMAC Stiffness Score (2 questions about stiffness where: 0=no stiffness to 10=extreme stiffness) for a total possible Index Score of 0 (best) to 240 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 8
Population: Safety population included all treated participants based on the actual treatment received.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 61 | 60
Score on a scale
  Baseline | 104.5 (36.53) | 107.6 (37.44)
  Change from Baseline at Week 8 (n=59,59) | -46.5 (35.21) | -43.8 (47.25)

3. Secondary Outcome: Change From Baseline in WOMAC Pain Score
Description: The WOMAC Pain Score included 5 questions about pain where: 0=no pain to 10=extreme pain for a total possible score of 0 (best) to 50 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 8
Population: Safety population included all treated participants based on the actual treatment received.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 61 | 60
Score on a scale
  Baseline | 23.9 (6.76) | 24.3 (7.01)
  Change from Baseline at Week 8 (n=59,59) | -10.7 (7.27) | -11.0 (9.75)

4. Secondary Outcome: Change From Baseline in WOMAC Physical Function Score
Description: The WOMAC Physical Function Score included 17 questions about the difficulty of daily activities where: 0=no difficulty to 10=extreme difficulty for a total possible score of 0 (best) to 170 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 8
Population: Safety population included all treated participants based on the actual treatment received.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 61 | 60
Score on a scale
  Baseline | 71.0 (28.43) | 73.3 (29.77)
  Change from Baseline at Week 8 (n=59,59 ) | -31.7 (26.41) | -28.6 (35.26)

5. Secondary Outcome: Patient Global Impression of Change Score
Description: The participants rated the change in their health status since enrollment using a 7-point scale where: +3=very much improved, +2=much improved, +1=minimally improved, 0=no change, -1=minimally worse, -2=much worse and -3=very much worse. Negative scores indicated worsening and positive scores indicated improvement.
Time Frame: Week 8
Population: Participants from the Safety population (all treated participants based on the actual treatment received) with data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 59 | 59
Score on a scale | 1.3 (1.28) | 1.0 (1.38)

6. Primary Outcome: Change From Baseline in the Average Daily Worst Pain Intensity Score at Week 8
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: Safety population included all treated participants based on the actual treatment received.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 61 | 60
Score on a scale
  Baseline | 6.4 (1.09) | 6.5 (1.28)
  Change from Baseline at Week 8 | -2.2 (1.96) | -2.3 (2.15)

7. Primary Outcome: Change From Baseline in the Average Daily Worst Pain Intensity Score at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Safety population included all treated participants based on the actual treatment received.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 61 | 60
Score on a scale
  Baseline | 6.4 (1.09) | 6.5 (1.28)
  Change from Baseline at Week 12 | -2.2 (1.97) | -2.5 (2.24)

8. Post Hoc Outcome: Change From Baseline in the Average Daily Worst Pain Intensity Score in the Nociceptive Pain Group
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8 and 12
Population: Participants from the Safety population (all treated participants based on the actual treatment received) in a subgroup of patients with nociceptive pain (pain that is caused by nerves that react to injury or damage) at Baseline.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 36 | 32
Score on a scale
  Baseline | 6.4 (1.01) | 6.4 (1.35)
  Change from Baseline at Week 4 | -1.9 (1.56) | -1.5 (1.58)
  Change from Baseline at Week 8 | -2.6 (2.01) | -1.8 (2.01)
  Change from Baseline at Week 12 | -2.6 (1.79) | -2.0 (2.27)

9. Post Hoc Outcome: Change From Baseline in WOMAC Pain Score in the Nociceptive Pain Group
Description: as for outcome 3
Time Frame: Baseline, Week 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 36 | 32
Score on a scale
  Baseline | 22.7 (5.95) | 22.9 (6.98)
  Change from Baseline at Week 8 (n=35,31) | -11.0 (7.09) | -7.5 (9.00)

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Type A | Placebo
Serious Adverse Events (participants affected / at risk) | 1/61 | 0/60
Other Adverse Events (participants affected / at risk) | 7/61 | 14/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=61) | Placebo (N=60)
Cerebrovascular accident (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=61) | Placebo (N=60)
Nasopharyngitis (Infections and infestations) | 1 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.